CLINICAL TRIAL: NCT02883998
Title: Formal vs. Home-Based Physical Therapy After Unicompartmental Knee
Brief Title: Formal vs. Home-Based Physical Therapy After Unicompartmental Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Rothman Institute Orthopaedics (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16021505
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis
Keywords: home-based physical therapy; outpatient physical therapy; unicompartmental knee arthroplasty; PT (Physical Therapy); osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient Physical Therapy Group (Active Comparator): Once the patient is cleared for discharged from the hospital, the patient will be given a prescription for outpatient physical therapy to attend 3 times per week for 6 weeks.
  Interventions: Other: Outpatient Physical Therapy
- Home Base Physical Therapy Group (Experimental): Patients will be provided a packet of exercises and equipment to perform the home based physical therapy program. Patients will attend a single session of outpatient physical therapy prior to surgery no more than 4 weeks prior to the procedure to teach the patient how to perform the exercises.
  Interventions: Other: Home Base Physical Therapy

INTERVENTIONS:
Other: Outpatient Physical Therapy — traditional outpatient physical therapy which occurs at a physical therapy office
  Arms: Outpatient Physical Therapy Group
Other: Home Base Physical Therapy — Patients will be provided a packet of exercises via a website which allows access to instructional physical therapy videos specifically designated for UKA patients and equipment to perform the home based physical therapy
  Arms: Home Base Physical Therapy Group

SUMMARY:
To determine whether home-based physical therapy (HBPT) is not clinically inferior to formal outpatient physical therapy (OPT) after hospital discharge of patients undergoing a unicompartmental knee arthroplasty (UKA).

DETAILED DESCRIPTION:
Given that current practice trends are requiring treatments to be both clinically and cost effective, research has begun to focus on evaluating the effect of specific interventions. Many surgeon and patients have believed formal OPT is necessary to optimize functional outcomes following orthopaedic procedures. However, the literature has begun to call into question the need for OPT following total hip arthroplasty, total knee arthroplasty, total shoulder arthroplasty, anterior cruciate ligament reconstruction, meniscectomy, and rotator cuff repair.

A randomized controlled trial was done to compare face-to-face rehabilitation with in-home telerehabilitation following total knee arthroplasty. Utilizing the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) as the primary outcome, the authors demonstrated noninferiority of telerehabilitation compared to face-to-face rehabilitation. Other secondary outcomes of Knee Injury and Osteoarthritis Outcome Score (KOOS), range of motion, and isometric strength did not exhibit a difference between the treatment groups. (see citation below)

Based on these findings, it appears that the high cost of formal OPT doesn't translate into a meaningful improvement of functional outcome. Because patient's undergoing UKA have a higher pre-operative functional status than patients having a TKA (Total Knee Arthroplasty), it is reasonable to think that patients following a UKA are better equipped to succeed with HBPT. As a result, the hypothesis of the current study is that HBPT will prove to be non-inferior to formal OPT in the setting of UKA.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a unicompartmental knee arthroplasty

Exclusion Criteria:

* Require inpatient physical therapy beyond post-operative day one
* < 18 years old
* Decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Knee Society Score | at 3 weeks, 3 months, and 1 year after surgery
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index | at 3 weeks, 3 months, and 1 year after surgery
Change from baseline in Knee range of motion | at 3 weeks, 3 months, and 1 year after surgery

SECONDARY OUTCOMES:
Complications | Will be assessed at 3 weeks, 3 months, and 1 year after surgery
  Deep Vein Thrombosis or Pulmonary Embolus Return to the OR within 30 days Re-admission within 30 days Superficial infection Deep infection Periprosthetic fracture Knee stiffness (defined as < 90 degrees flexion at 3 weeks post-operative or < 110 degrees flexion at 6 weeks post-operative)
Cost comparison | Will be assessed at 3 weeks, 3 months, and 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Craig Della Valle, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moffet H, Tousignant M, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Ranger P, Belzile EL, Dimentberg R. In-Home Telerehabilitation Compared with Face-to-Face Rehabilitation After Total Knee Arthroplasty: A Noninferiority Randomized Controlled Trial. J Bone Joint Surg Am. 2015 Jul 15;97(14):1129-41. doi: 10.2106/JBJS.N.01066. PMID 26178888